CLINICAL TRIAL: NCT04279379
Title: Combination of Sintilimab and Decitabine for Patients With Relapsed/Refractory or Advanced NK/T-cell Lymphoma : a Single Arm,Open-lable,Phase II Study
Brief Title: Sintilimab and Decitabine for Patients With Relapsed/Refractory or Advanced NK/T-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, JING-WEN WANG, Director of department of hematology, Beijing Tongren Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRhos-ENKTCL-2
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Extranodal NK/T-cell Lymphoma
Keywords: extranodal NK/T-cell lymphoma; PD-1 blockade; decitabine; sintilimab; hypomethylation; epigenetics
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — sintilimab; spartalizumab; Decitabine

STUDY DESIGN:
Intervention Model Description: treatment with sintilimab and decitabine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): Sintilimab,200mg,ivdrip,day1 Decitabine 10mg d1-5, ivdrip, repeated every 3 weeks.
  Interventions: Drug: Sintilimab; Drug: Decitabine

INTERVENTIONS:
Drug: Sintilimab — 200mg d1,ivdrip, repeated every 3 weeks
  Other Names: anti-PD-1-antibody
Drug: Decitabine — 10mg d1-5, ivdrip,repeated every 3 weeks
  Other Names: hypomethylating agents

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Sintilimab in combination with decitabine in the treatment of Relapsed/Refractory or advanced NK/T-cell lymphoma patients

DETAILED DESCRIPTION:
Previous study has confirmed the efficacy of anti-PD-1 antibodies (including pembrolizumab or sintilimab). However, the CR rate of PD-1 antibody monotherapy is too low. Previous studies have demonstrated that decitabine may activate the T cells and enhance the efficacy of PD-1 antibodies in Hodgkin Lymphoma. Thus, the investigators aim to evaluate the efficacy and safety of sintilimab in combination with decitabine in the treatment of NK/T cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

Histopathology and immunohistochemistry confirmed diagnosis of NK/Tcell lymphoma according to WHO 2016 criteria.

* refractory or relapsed after initial remission, or stage III-IV de novo patients
* PET/CT or CT/MRI with at least one objectively evaluable lesion.
* General status ECOG score 0-3 points.
* The laboratory test within 1 week before enrollment meets the following conditions: Blood routine: Hb>80g/L, PLT>50×10e9/L. Liver function: ALT, AST, TBIL ≤2 times the upper limit of normal. Renal function: Cr is normal. Cardiac function: LVEF≥50%, ECG does not suggest any acute myocardial infarction, arrhythmia or atrioventricular conduction above I Blocking.
* Sign the informed consent form

Exclusion Criteria:

Active infection requires ICU treatment. Concomitant HIV infection or active infection with HBV, HCV. Patients who are infected with HBV but not active hepatitis at the same time are notexcluded.

Significant organ dysfunction Pregnant and lactating women. Had a history of autoimmune diseases, and disease was active in the last 6 months.

Those who were known to be allergic to drugs in the study regimen. Patients with other tumors who require surgery or chemotherapy within 6 months.

• Other experimental drugs are being used.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
complete response rate | 24 weeks ±7 days
  evaluated by PET-CT and MRI, according to Lugano 2014 criteria

SECONDARY OUTCOMES:
overall response rate | 24 weeks ±7 days
  evaluated by PET-CT and MRI, according to Lugano 2014 criteria
1-year progression free survival rate | up to 1year after enrollment
  time from date of enrollment to date of disease progression, death of any reason, whichever comes first
1-year overall survival rate | up to 1year after enrollment
  time from date of enrollment to date death of any reason

CONTACTS AND LOCATIONS:
Overall Officials: Jing-wen Wang, M.D., Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No